CLINICAL TRIAL: NCT04068649
Title: A Phase 2 Randomized Study With a Non-randomized Cohort : Assessing Single-Fraction SBRT Versus Standard Palliative Radiation in Patients With Metastatic Disease (ASTEROID)
Brief Title: Single-Fraction SBRT Versus Standard Palliative Radiation Therapy in Treating Patients With Metastatic Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Roswell Park Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: I 81318; NCI-2019-04859 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); I 81318 (Other: Roswell Park Cancer Institute)
Record Dates: First submitted 2019-08-21; First posted 2019-08-28 (Actual); Last update posted 2025-04-25 (Actual); Status verified 2025-04

CONDITIONS: Metastatic Malignant Neoplasm
MeSH Terms: conditions — Neoplasm Metastasis | interventions — Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Arm I (palliative RT) (Experimental): Patients undergo 1, 3-5, 5-6, or 10 fractions of palliative RT deemed appropriate by the treating physician.
  Interventions: Radiation: Palliative Radiation Therapy; Other: Quality-of-Life Assessment; Other: Questionnaire Administration
- Arm II (SBRT) (Experimental): Patients undergo single fraction SBRT.
  Interventions: Other: Quality-of-Life Assessment; Other: Questionnaire Administration; Radiation: Stereotactic Body Radiation Therapy

INTERVENTIONS:
Radiation: Palliative Radiation Therapy — Undergo palliative RT
  Arms: Arm I (palliative RT)
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies
Radiation: Stereotactic Body Radiation Therapy — Undergo SBRT
  Other Names: SABR; SBRT; Stereotactic Ablative Body Radiation Therapy
  Arms: Arm II (SBRT)

SUMMARY:
This phase II trial studies how well single-fraction stereotactic body radiation therapy (SBRT) works when compared to standard radiation therapy in treating patients with cancer that has spread to other places in the body (metastatic). Stereotactic body radiation therapy uses special equipment to position a patient and deliver radiation to tumors with high precision. This method can kill tumor cells with fewer doses over a shorter period and cause less damage to normal tissue.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess patient-reported pain response and quality of life (QoL) in patients randomized to either single-fraction stereotactic body radiation therapy (SBRT) or non-SBRT palliative radiation therapy for metastatic disease.

SECONDARY OBJECTIVES:

I. Compare overall survival for patients undergoing single fraction SBRT versus non-SBRT palliative radiation therapy.

EXPLORATORY OBJECTIVES:

I. Assess for changes in immune markers. II. Assess toxicity related to radiation treatment. III. Assess change in frailty index and cognitive function over time in patients undergoing treatment for metastatic cancer.

IV. Evaluate the effect of circadian rhythm and radiation treatment time on outcomes.

V. Assess the utility of the Pain Catastrophizing Index in patients undergoing radiation treatment for metastatic cancer.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM I: Patients undergo 1, 3-5, 5-6, or 10 fractions of palliative radiation therapy (RT) deemed appropriate by the treating physician.

ARM II: Patients undergo single fraction SBRT.

After completion of study treatment, patients may be followed up at 5 and 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed malignancy
* Clinical or pathologic evidence of metastatic disease
* A site of malignant disease causing symptoms, or for which symptoms are imminent, in which radiation may be used for relief or prophylaxis
* Participants of child-bearing potential must agree to use adequate contraceptive methods (e.g., hormonal or barrier method of birth control; abstinence) prior to study entry. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately
* Participants with synchronous primary malignancies must have either: 1) documented control of their second malignancy or 2) have pathological confirmation of the metastatic lesion/disease site being targeted
* Participant must be willing and able to participate in protocol requirements, including pre- and post-treatment survey evaluations and clinical assessments
* Participant must understand the investigational nature of this study and sign an Independent Ethics Committee/Institutional Review Board approved written informed consent form prior to receiving any study related procedure

Exclusion Criteria:

* Prior radiation therapy targeting the same area for which radiation treatment is being planned (i.e., re-irradiation to a specific site of metastatic disease)
* Participants with known brain metastases
* Pregnant or nursing female participants
* Participants who are unable to accurately or reliably recount their pain medication regimens, including type, amount, or frequency of pain medication usage
* Participants who require or are being planned for surgical stabilization or metastasectomy of the planned radiation site
* Severe, active co-morbidity defined as follows:

  * Unstable angina and/or congestive heart failure requiring hospitalization within the last 3 months;
  * Transmural myocardial infarction within the last 3 months;
  * Acute bacterial or fungal infection requiring intravenous antibiotics at the time of registration;
  * Chronic obstructive pulmonary disease exacerbation or other respiratory illness requiring hospitalization or precluding study therapy at the time of registration
* Unwilling or unable to follow protocol requirements
* Any condition which, in the investigator?s opinion, deems the patient unable to participate in enrollment
* Adults unable to consent
* Individuals who are not yet adults (infants, children, teenagers)
* Pregnant women
* Prisoners

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1500 (Estimated)
Dates: Start 2019-11-18 (Actual); Primary Completion 2027-11-18 (Estimated); Study Completion 2027-11-18 (Estimated)

PRIMARY OUTCOMES:
Pain responses | Baseline up to 12 weeks
  Will be quantified using the pain scales from the Brief Pain Inventory (BPI). Will be an analysis-of-covariance.
Change in Quality of life | Baseline up to 12 weeks
  Will be measured with European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Core 30. Will be an analysis-of-covariance.

SECONDARY OUTCOMES:
Overall survival | Up to date of last follow-up or date of death, at the time of study analysis, assessed up to 12 weeks
  Will be assessed by chart review. Will be carried out using a Cox proportional hazards regression model.

OTHER OUTCOMES:
Changes in immune markers | Up to 12 weeks
  Changes in the mediators of tumor antigen presentation, costimulatory molecules, immune effector cell populations, such as CD4+ and CD8+ T-cells, T regulatory cells (CD4+CD25+FoxP3+), natural killer cells, monocytes, macrophages, dendritic cells and myeloid derived suppressor cells will be assessed.
Hospitalization resulting from radiation treatment | Up to 12 weeks
  Will be recorded. Any acute (=< 180 days after the end of radiation therapy [RT]) and late (> 180 days after the end of RT) toxicities will be documented using the Cancer Therapy Evaluation Program National Cancer Institute Common Terminology Criteria for Adverse Events version 5.0.
Cognitive function | Up to 12 weeks
  Will be measured using combined G8 questionnaire and Montreal Cognitive Assessment assessments.
Pain catastrophizing scale | Up to 12 weeks
  Will be measured in conjunction with pain endpoints.
Impact of the time of day of treatment on patient outcomes | Up to 12 weeks
  A retrospective analysis will be used.
Frailty Assessment | Up to 12 weeks
  Frailty will be determined using the Fried Frailty Index

CONTACTS AND LOCATIONS:
Overall Officials: Anurag K Singh, Principal Investigator — Roswell Park Cancer Institute
Locations (3):
- United States (3):
  - Roswell Park Cancer Institute, Buffalo, New York
  - The Cancer Institute at St. Francis Hospital, East Hills, New York
  - Good Samaritan Hospital, West Islip, New York